CLINICAL TRIAL: NCT04193332
Title: Near Infrared (NIR) Autofluorescence Image-guided Thyroid Surgery Can Prevent Post-thyroidectomy Hypoparathyroidism
Brief Title: Near Infrared (NIR) Autofluorescence Image-guided Thyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Cluster for molecular imaging, Denmark (Unknown); Dept of Otorhinolaryngology and Maxillofacial Surgery, Zealand University Hospital, Denmark (Unknown)
Responsible Party: Principal Investigator, Eva Lykke, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H19010211
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Hypoparathyroidism Postprocedural; Hypocalcemia; Surgery--Complications
Keywords: thyroide surgery; total thyroidectomy; compltion thyroidectomy; parathyroidectomy; autofluorescense; NIR; near-infrared; optical imaging
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plus NIR optical imaging (Experimental): NIR optical imaging assisted identification of parathyroid glands during thyroid surgery
  Interventions: Device: NIR optical imaging camera
- Minus NIR optical imaging (No Intervention): Conventional identification of parathyroid glands during thyroid surgery

INTERVENTIONS:
Device: NIR optical imaging camera — NIR optical imaging assisted identification of parathyroid glands during thyroid surgery using parathyroid gland autofluorescense
  Arms: Plus NIR optical imaging

SUMMARY:
The objective of this ongoing randomized controlled trial is to examine whether the use of intra-operative NIR(near infrared) camera can reduce the number of patients who experience transient or persistent hypoparathyroidism after total thyroidectomy and completion thyroidectomy, both in malignant and benign thyroid disease.

DETAILED DESCRIPTION:
Patients admitted to total thyroidectomy or completion thyroidectomy is ramdomized to:

1. Intervention: NIR optic imaging assisted identification of the parathyroid glands during thyroidectomy using parathyroid gland autofluorescence.
2. Control: Conventional thyroidectomy and parathyroid identification by the surgeon.

Measurements:

PTH and ionized-Ca blood samples are collected preoperatively, within 12 hours postoperatively and at 1-, 3-, 9- and 12-months follow-up.

Anticipated 214 patients are included, all of which participate in 3 months follow-up. Only patients with persistent hypoparathyroidism at this point continue til maximum 12 months follow-up.

An interim analysis will be conducted when inclusion of anticipated 128 patients and 3 months follow-up is reached.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand patient information and to give written informed consent
* Patients admitted to either total thyroidectomy og completion thyroidectomy, both benign and malign.

Exclusion Criteria:

* Not able to understand patient information and to give written informed consent
* Previous parathyroid surgery or other parathyroid decease
* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2019-08-16 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative hypoparathyroidism | 24 months-follow-up
  Hypoparathyroidism defined as: PTH < 1,6 pmol/L and based on European Society of Endocrinology Clinical Guideline

SECONDARY OUTCOMES:
Postoperative hypocalcemia | 12 months follow-up
  Hypocalcemia defined as: ionized Calcium < 1,15 mmol/L
Time | Immediately after surgery
  Duration of surgery
Parathyroidglands identified by NIR light | During surgery
  Number of identified by NIR light vs. white light

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Buchwald, MDSc, PhD, Study Director — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Dept of Otorhinolaryngology and Maxillofacial Surgery, Zealand University Hospital, Denmark, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbaci M, De Leeuw F, Breuskin I, Casiraghi O, Lakhdar AB, Ghanem W, Laplace-Builhe C, Hartl D. Parathyroid gland management using optical technologies during thyroidectomy or parathyroidectomy: A systematic review. Oral Oncol. 2018 Dec;87:186-196. doi: 10.1016/j.oraloncology.2018.11.011. Epub 2018 Nov 16. PMID 30527238
- [Background] Dip F, Falco J, Verna S, Prunello M, Loccisano M, Quadri P, White K, Rosenthal R. Randomized Controlled Trial Comparing White Light with Near-Infrared Autofluorescence for Parathyroid Gland Identification During Total Thyroidectomy. J Am Coll Surg. 2019 May;228(5):744-751. doi: 10.1016/j.jamcollsurg.2018.12.044. Epub 2019 Jan 31. PMID 30710614
- [Background] Benmiloud F, Rebaudet S, Varoquaux A, Penaranda G, Bannier M, Denizot A. Impact of autofluorescence-based identification of parathyroids during total thyroidectomy on postoperative hypocalcemia: a before and after controlled study. Surgery. 2018 Jan;163(1):23-30. doi: 10.1016/j.surg.2017.06.022. Epub 2017 Nov 6. PMID 29122325
- [Derived] Lykke E, Christensen A, Juhl K, Feldt-Rasmussen U, Friberg Hitz M, Svenningsen Sjostedt SM, Holst Hahn C, Kraik Svensson DM, Kanstrup Springborg K, Stage MG, Bjorn Hvilsom G, Hilsted LM, Dahl M, Lelkaitis G, Kjaer A, Homoe P, von Buchwald C. Effect of near infrared autofluorescence guided total thyroidectomy on postoperative hypoparathyroidism: a randomized clinical trial. Eur Arch Otorhinolaryngol. 2023 May;280(5):2593-2603. doi: 10.1007/s00405-023-07867-4. Epub 2023 Feb 28. PMID 36853388